CLINICAL TRIAL: NCT05820373
Title: The Effect of Yoga Therapy on Post-operative Side-effects Among Women With Breast Cancer: a Randomized Controlled Trial
Brief Title: The Effect of Yoga Therapy on Post-operative Side-effects Among Women With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: hong Kong Cancer Fund (Unknown)
Responsible Party: Principal Investigator, Wendy Wing Tak Lam, Associate professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Yoga2013
Record Dates: First submitted 2023-03-15; First posted 2023-04-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer; Yoga Therapy; Shoulder Joint Motion; Scar Contracture
Keywords: Yoga therapy; Breast Cancer; scar contracture; shoulder joint motion
MeSH Terms: conditions — Breast Neoplasms | interventions — Yoga

STUDY DESIGN:
Intervention Model Description: The investigators will use a block randomization structure with randomly permuted block sizes of 2, 4 and 6 to ensure a close balance of the numbers in each arm. Randomization (by a statistician) occurs prior to eligible patients attending the clinic to minimize opportunities for selection bias.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigator, care provider, and outcomes assessor are masked in terms of not knowing to which condition the participants will be randomized until after the completion of the baseline assessment. The outcomes assessor will break the envelope for the next eligible participant and inform them the allocation result.
  The participants are masked in terms of not knowing that the yoga therapy is hypothesized to yield larger effects than the others.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group (Experimental): Women being allocated to the intervention group will attend a 12-week, bi-weekly, specially designed yoga therapy course.
  Interventions: Behavioral: Yoga therapy
- Active control group (Active Comparator): Women being allocated to the active control group will attend a 12-week, weekly, relaxation course.
  Interventions: Behavioral: Active control group
- Passive control group (Placebo Comparator): The passive control intervention will be the standard post-operative exercises which are currently introduced to women following surgery, for all women allocated to the control group.
  Interventions: Behavioral: Passive control group

INTERVENTIONS:
Behavioral: Yoga therapy — Women being allocated to the intervention group will attend a 12-week, bi-weekly, specially designed yoga therapy course. In each yoga class, participants will be taught to perform a standardized yoga sequence including postures and breathing exercise. Each class lasts 60 minutes. A DVD demonstrating the yoga sequence will be given to each participant to prompt daily home practice.
  Arms: Intervention group
Behavioral: Active control group — Women being allocated to the active control group will attend a 12-week, weekly, relaxation course. In each relaxation class, participants will be taught to learn mediation and guided relaxation, called Shavasana. Participants will be asked to lie on their back, with legs apart and their eyes closed. During the practice, participants learn how to relax the body and breath normally. Each session lasts 60 minutes.
  Arms: Active control group
Behavioral: Passive control group — The passtive control intervention will be the standard post-operative exercises which are currently introduced to women following surgery, for all women allocated to the control group. A DVD demonstrating the post-operative exercise will be given to participants to practice at home daily.
  Arms: Passive control group

SUMMARY:
The present study evaluates the effect of yoga therapy on scarring contractures and shoulder joint motion and range in women diagnosed with breast cancer. A single-blinded prospective, randomized controlled trial will be used.

DETAILED DESCRIPTION:
To conduct a study to evaluate the effect of yoga therapy on scarring contractures and shoulder joint motion and range in women diagnosed with breast cancer using a single-blinded prospective, randomized controlled trial.

The aims are to test:

1. To evaluate the impact of yoga therapy on scarring contractures and range of motion in shoulder joints among women recovering from surgical treatment of breast cancer.
2. To evaluate the impact of yoga therapy on health-related quality of life and symptom distress.

Primary Hypotheses

1. Intervention and control groups mean scores on measures of shoulder movement range will show no differences at baseline or significant changes at the immediate post-intervention, 3rd, 6th, and 12th month post-intervention.
2. Mean scores of quality of life and symptom distress between intervention and control groups at the immediate post-intervention, 3rd, 6th, and 12th month post-intervention will show no differences relative to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Cantonese-speaking Chinese patients
* were newly diagnosed with breast cancer
* had completed breast cancer surgery plus chemotherapy
* were able to give consent

Exclusion Criteria:

* Patients who have residual breast tumors or loco-regional metastasis after treatment
* who were practicing yoga since the diagnosis of breast cancer
* or are otherwise physically unable to yoga

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female breast cancer patients were eligible to the present study
Enrollment: 444 (Actual)
Dates: Start 2013-05-14 (Actual); Primary Completion 2018-11-29 (Actual); Study Completion 2018-11-29 (Actual)

PRIMARY OUTCOMES:
Change in shoulder rotation flexibility | Baseline, immediate post-intervention, 3rd, 6th, and 12th month post-intervention.
  Start by holding a strap in front of the body with both hands wide apart and palms facing downwards. Lift the strap over the head to behind the back, maintaining the hand grip on the object. This movement must be made with extended arms. Repeat the movement, moving hands closer together each time until the movement cannot be completed with straight arms. To assess the flexibility, the best score of three trials is recorded. The score is the angle of fanning out, in degrees, calculated with the formula S/2L, where S = how much the sliding handle shifted in cm during the movement; L = length of arm in cm from acromion to the metacarpophalangeal joint of the middle finger.
Change in shoulder range of motion | Baseline, immediate post-intervention, 3rd, 6th, and 12th month post-intervention.
  Back scratch test. This test is performed in the standing position. Place one hand behind the head and back over the shoulder, then reach as far as possible down the middle of the back, with the palm touching the body and the fingers directed downwards. Place the other arm behind the back, palm facing outward and fingers upward and reach up as far as possible attempting to touch or overlap the middle fingers of both hands. To assess the range of motion, measure the distance between the tips of the middle fingers. If the fingertips touch then the score is zero. If they do not touch, measure the distance between the finger tips (i.e. a negative score). If they overlap, measure by how much (i.e. a positive score). Take two measures and use the best score.

SECONDARY OUTCOMES:
Change in generic quality of life | Baseline, immediate post-intervention, 3rd, 6th, and 12th month post-intervention.
  The Standard Chinese version of the European Organization Research Treatment Cancer (EORTC) general quality of life questionnaire (QLQ-C30) is used to assess health-related quality of life. The EORTC QLQ-C30 includes 30 items that measure five function scales (physical, role, emotional, cognitive, and social), three symptom scales (fatigue, pain, and nausea/vomiting), a global health QoL subscale, five single symptom items (dyspnea, appetite loss, sleep disturbance, constipation, and diarrhea) and financial difficulty. A 4-point Likert scale ranging from 0 "Not at all" to 3 "Very much" is used. All the subscales range from 0 to 100. Higher scores on the subscales of function, global health status, and symptoms indicate healthy levels of functioning, better quality of life, and higher levels of symptomatology or problems, respectively.
Change in the severity of pain | Baseline, immediate post-intervention, 3rd, 6th, and 12th month post-intervention.
  The severity of current pain and pain over the previous 6 months is assessed using the Chronic Pain Grade questionnaire. Patients are asked about the severity, site, and duration of their pain. All items are scored on an 11-point Likert scale, with responses ranging from 0-10. Scores are calculated for 3 subscales: the characteristic pain intensity score, which ranges from 0-100, is calculated as the mean intensity ratings for reported current, worst, and average pain; the disability score, which ranges from 0-100, is calculated as the mean rating for difficulty performing daily, social, and work activities; and the disability points score, which ranges from 0-3, is derived from a combination of ranked categories of number of disability days and disability score. Higher scores indicates higher levels of pain intensity, greater difficulty performing daily, social, and work activities, and greater disability, respectively.
Change in psychological distress | Baseline, immediate post-intervention, 3rd, 6th, and 12th month post-intervention.
  The 14-item Hospital Anxiety and Depression Scale (HADS) measures anxiety and depression. Respondents will be asked to rate each of the 14 statements using a 4-point scale to indicate how they have felt in the past week. Total scores for each subscale (7 items) range from 0 to 21, with higher scores indicating greater distress. This measure has been widely used in studies of cancer patients and has demonstrated good validity and reliability.
Change in quality of life (Breast cancer specific) | Baseline, immediate post-intervention, 3rd, 6th, and 12th month post-intervention.
  The Standard Chinese version of the breast cancer specific module of the European Organization Research Treatment Cancer (EORTC) quality of life questionnaire (QLQ- BR23) assesses health-related quality of life. The QLQ- BR23 is a breast cancer specific measure consisted of 23 items assessing four functional domains (body image, sexual functioning, sexual enjoyment, and future perspective) and four symptom scales (arm symptoms, breast symptoms, side effects of systemic therapy, and being upset by hair loss). A 4-point Likert scale ranging from 0 "Not at all" to 3 "Very much" is used. All the subscales range from 0 to 100. Higher scores on the subscales of function and symptoms indicate healthy levels of functioning and higher levels of symptomatology or problems, respectively.
Change in sleep quality | Baseline, immediate post-intervention, 3rd, 6th, and 12th month post-intervention.
  The 19-item Chinese version of the Pittsburgh Sleep Quality Index (PSQI) measures 7 components of sleep quality: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleep medication, and daytime dysfunction, in which each component scored from 0-3, with the global score ranging from 0-21. Higher scores indicate poorer sleep quality.
Change in fatigue | Baseline, immediate post-intervention, 3rd, 6th, and 12th month post-intervention.
  Fatigue is assessed using the Chalder Fatigue scale. The Chalder Fatigue scale is a 11-items scale measuring severity of physical and mental fatigue. Total fatigue score is obtained by summing all items, which are rated on a four-point Likert scale (0=not at all; 3=much more than usual). Higher scores indicate greater fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Wing Tak Lam, PhD, Principal Investigator — School of Public Health, The University of Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be available from the PI upon reasonable request.
Supporting Information: Study Protocol
Time Frame: Starting 6 months after publication
Access Criteria: Information will be available from the PI upon reasonable request. The author to review requests is the PI.